CLINICAL TRIAL: NCT02381535
Title: A Phase I Trial of AT13387 in Patients With Locoregionally Advanced Squamous Cell Carcinoma of the Head and Neck (LA-SCCHN) Receiving Concurrent Radiation and Cisplatin
Brief Title: Onalespib in Treating Patients With Locoregionally Advanced Squamous Cell Carcinoma of the Head and Neck Receiving Radiation Therapy and Cisplatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00256; NCI-2015-00256 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PJC-017; 9874 (Other: University Health Network Princess Margaret Cancer Center LAO); 9874 (Other: CTEP); UM1CA186644 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Stage III Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage III Laryngeal Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVA Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVB Oropharyngeal Squamous Cell Carcinoma AJCC v7
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiotherapy, Intensity-Modulated; (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (onalespib, cisplatin, IMRT) (Experimental): Patient receive onalespib IV over 1 hour on days -7, 3, 10, 24, 31, and 38 and cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, 36 and 43. Patients also undergo IMRT QD, 5 days a week over 7 weeks for a total of 35 fractions. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Onalespib; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Onalespib — Given IV
  Other Names: AT 13387; AT-13387; AT13387
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of onalespib when given together with intensity-modulated radiation therapy (IMRT) and cisplatin in treating patients with squamous cell carcinoma of the head and neck that has spread from where it started to nearby tissue or lymph nodes. Onalespib works by blocking a protein called HSP90. HSP90 helps protect cells from stress and supports many other proteins that cause cell growth. When HSP90 is blocked, tumor cell growth may be slowed or stopped and may die more easily when treated with chemotherapy and radiation. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. IMRT is a specialized radiation therapy that delivers beams of radiation of different intensities aimed at the tumor from many angles and may kill more tumor cells and cause less damage to normal tissue. Giving onalespib with cisplatin and IMRT may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and recommended phase II dose (RP2D) of onalespib (AT13387) in combination with concurrent cisplatin and radiotherapy in patients with locoregionally advanced squamous cell carcinoma of the head and neck (LA-SCCHN). (Dose Escalation Phase) II. To preliminarily evaluate the safety and preliminary efficacy of AT13387 in combination with concurrent cisplatin and radiotherapy in patients with LA-SCCHN. (Dose Expansion Phase)

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of AT13387 in combination with cisplatin and radiotherapy.

II. To evaluate the pharmacokinetics of cisplatin in combination with AT13387 and radiotherapy.

III. To assess for pharmacodynamics biomarkers for proof-of-mechanism. IIV. To assess for potential predictive biomarkers of efficacy. V. To document the toxicities associated with the administration of AT13387 in combination with cisplatin and radiotherapy in patients with LA-SCCHN.

VI. To explore and characterize predictive biomarkers for individual cancer patients utilizing genomic sequencing technologies.

VII. To provide preliminary disease-free survival, locoregional control, distant metastases-free survival, and overall survival.

OUTLINE: This is a dose-escalation study of onalespib.

Patients receive onalespib intravenously (IV) over 1 hour on days -7, 3, 10, 24, 31, and 38 and cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, 36, and 43. Patients also undergo IMRT once daily (QD), 5 days a week over 7 weeks for a total of 35 fractions. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 8 weeks, every 3 months for 1 year, and then every 6 months for 1 year. Beyond the first 2 years, patients may be followed up every 6 months for up to 3 years per institutional standards.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed, previously untreated squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx
* Tumors must be staged T1-4, N2b-3, M0 (human papillomavirus positive [HPV]+ or HPV negative [-]); patients with HPV+ tumors should have at least one high risk feature such as T4, N3, or smoking history of > 10 pack years
* The disease must be considered to be potentially curable by combined radiotherapy and cisplatin based chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 6 months
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets >= 100 x 10^9/L
* Serum creatinine =< 1.5 mg/dL (=< 120 umol/L) OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min
* Bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 2.5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN
* Proteinuria =< +1 on dipstick or =< 1 gram/24 hours
* Corrected QT using the Fridericia formula (QTcF) < 470 msec
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study participation, and for three months after the last dose of the drug; women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to registration and agree to use effective contraception throughout the treatment period and for 3 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception; males should avoid fathering children during and for at least three months after therapy is completed
* Ability to understand and the willingness to sign a written informed consent document
* Available for long-term follow-up of their disease after treatment

Exclusion Criteria:

* Patients with nasopharyngeal, paranasal sinus, skin, or unknown primary site disease
* Presence of distance metastases (M1)
* History of another malignancy; exception: patients who have been disease-free for > 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies, are eligible; consult the Cancer Therapy Evaluation Program (CTEP) Medical Monitor if unsure whether second malignancies meet the requirements specified above
* Previous head and neck radiation therapy
* Symptomatic peripheral neuropathy > grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) criteria
* Clinically significant sensorineural hearing impairment which may be worsened via cisplatin exposure (audiometric abnormalities without corresponding clinical deafness are not grounds for exclusion)
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to AT13387
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited: the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], ginkgo biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* History or current evidence/risk of visual loss syndromes, including but not limited to retinal vein occlusion (RVO), retinal detachment, macular degeneration, or visual migraine headaches
* History or evidence of cardiovascular risk including any of the following:

  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Patients with intra-cardiac defibrillators
* Known hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection are eligible); patients with known human immunodeficiency virus (HIV) infection are eligible if not on antiviral agents and cluster of differentiation (CD)4 counts are adequate (>= 500)
* HIV-positive patients on combination antiretroviral therapy are ineligible
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any condition or medical problem in addition to the underlying malignancy and organ dysfunction which the investigator feels would pose unacceptable risk
* Breastfeeding patients are ineligible

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by dose-limiting toxicity (DLT) of onalespib in combination with concurrent cisplatin and radiation therapy graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 | 8 weeks
Pharmacokinetic (PK) profile of onalespib in combination with cisplatin and radiation therapy | Baseline, 0.5, 1, 2, 3, 4, 6, 8, 9, and 24 hours on day -7; baseline, 0.5, 1, 2, 3, 4, 6, 8, 9, 24 hours on day 9; and baseline on day 24
  Attempts to model associations between pharmacokinetic data with toxicity profiles will be performed primarily using descriptive statistics; however, logistic regression may be used if warranted.
PK profile of cisplatin in combination with concurrent onalespib and radiotherapy | Baseline, at end of cisplatin infusion, at 2, 4, 6, and 8-9 on day 8, and 24 hours on day 9, and at baseline on days 22 and 29
  Attempts to model associations between pharmacokinetic data with toxicity profiles will be performed primarily using descriptive statistics; however, logistic regression may be used if warranted.

SECONDARY OUTCOMES:
Incidence of non-DLT adverse events (AEs) | Up to 2 years
  Frequency and severity of AEs will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest. AEs will be summarized using all AEs experienced, although a sub-analysis may be conducted including only those adverse events in which the treating physician deems possibly, probably or definitely attributable to one or both study treatments. Attempts to model associations between pharmacokinetic data with toxicity profiles will be performed primarily using descriptive statistics; however, logistic regression may be used if warranted.
Antitumor activity | Up to 2 years
  Predictors of clinical outcomes will be investigated using logistic regression, Cox proportional hazards regression and/or generalized estimating equations as appropriate. Potential predictors include clinical predictors and molecular correlates. Descriptive statistics and plotting of data will also be used to better understand potential relationships.
Predictive biomarkers for individual cancer patients utilizing biopsies and genomic sequencing technologies | Up to week 7

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Hope, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (2):
- Yale University, New Haven, Connecticut, United States
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada